CLINICAL TRIAL: NCT05392634
Title: Рrospective Multicenter Randomized 3 Phase Study Evaluating the Role of Prolonged Antibiotic Prophylaxis as a Measure to Reduce the Incidence of Postoperative Complications After Radical Cystectomy With ERAS Protocol
Brief Title: Multicentral Preventive Antibiotics With Cystectomy Within Enhanced Recovery After Surgery
Acronym: MACS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Collaborators: The Foundation for Cancer Research Support (RakFond) (Unknown)
Responsible Party: Principal Investigator, Berkut Mariya, Principal Investigator, N.N. Petrov National Medical Research Center of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MACS-1
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Bladder Cancer
Keywords: radical cystectomy; antibiotic prophylaxis; ERAS protocol; muscle-invasive bladder cancer; urinary diversion
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Meropenem; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin/ Cefuroksim (Active Comparator): standard antibiotic prophylaxis 24 hours
  Interventions: Drug: Amoxicillin+clavulanic acid 1200 mg or Cefuroksim 1500mg
- Meropenem (Experimental): preventive antibiotic therapy within 5 days from the date of the skin incision
  Interventions: Drug: Meropenem 1000 mg

INTERVENTIONS:
Drug: Meropenem 1000 mg — Group B: prolonged antibiotic prophylaxis >72 hours (5 days) from the moment of the skin incision in accordance with the selected clinic drug + correction of the appointment based on clinical events after 5 days.
  Arms: Meropenem
Drug: Amoxicillin+clavulanic acid 1200 mg or Cefuroksim 1500mg — Group A: antibiotic prophylaxis within 24 hours from the moment of skin incision according to local clinical practice;
  Arms: Amoxicillin/ Cefuroksim

SUMMARY:
The current usage of antibiotic prophylaxis (AP) in radical cystectomy (RC) is aimed to reducing the incidence of surgical site infections and incidence of unnecessary prescribing of antibiotics. There are a huge number of different AP protocols according to Urological Associations. However, there is no convincing evidence to support variations and duration of AP which requires a randomized clinical trial on AP when performing variants of RC with uroderivation.

Research hypothesis: The use of prolonged antibiotic prophylaxis (5 days), depending on the glomerular filtration rate, does not affect the incidence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of very high risk non muscle-invasive bladder carcinoma (cT1NoMo) or muscle-invasive bladder carcinoma (cT2-T4NxM0) with or without neoadjuvant therapy (chemotherapy or immunotherapy are both possible);
* patient should be eligible for radical cystectomy (RC) + pelvic lymph node dissection (PLND), and agreement to undergo curative intent standard RC + PLND (including prostatectomy or hysterectomy if applicable) according to surgeon opinion;
* pelvic lymph node dissection is engaged in two possible variants: extended level to intersection of ureter and iliac vessels; superextended level - up to aortic bifurcation;
* urinary diversion is engaged in two possible variants: orthotopic diversion (J- or U-pouch reservoirs), heterotopic diversion in the Mainz-I modification, Bricker;
* male or female is at least 18 years old at the time of signing the informed consent form;
* female patient is eligible to participate if she is not pregnant, not breastfeeding;
* ECOG performance status of 0 or 1;
* adequate organ function (in accordance with laboratory standards);
* used valid protocol for Enhanced Recovery After Surgery (ERAS protocol) at Hospital (oncourological department);

Exclusion Criteria:

* known additional non-urothelial malignancy that is progressing or has required active anticancer treatment ≤3 years of study randomization, with certain exceptions;
* diagnosis of immunodeficiency or receipt of chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug;
* replacement doses of corticosteroids are permitted for participants with adrenal insufficiency;
* evidences of uncontrolled diseases (diabetes mellites, noninfectious pneumonitis that required steroids, et.) or any conditions which interfere with the conduct of the research procedures according to doctor opinion;
* presence of 2 or more criteria for systemic inflammatory response syndrome (SIRS) at the time of the patient's admission to the hospital (assessment of these factors 3-7 days before randomization):

  * temperature ≥ 38˚С or ≤ 36˚С;
  * heart rate (HR) ≥ 90 / min;
  * respiratory rate < 20/min or hyperventilation (Pa CO2 ≤ 32 mm Hg);
  * blood leukocytes >12 ∙ 109 / l or < 4 ∙ 109 / l, or immature forms > 10%
* prohibited urinary diversion when planning surgery and signing voluntary consent: diversion into continuous intestine (ureterosigmostomy, Mainz-pouch II operation);
* inadequate organ function:

  * Neutrophils <1.5 x 10 ^ 9 / l
  * Platelets <100 x 10 ^ 9 / l
  * ALT> 3 x VGN
  * AST> 3 x VGN
  * Bilirubin> 1.5 x ULN
  * GFR level <35 ml / min

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Event rate | 90 days after Radical cystectomy
  Determine the frequency of events of clinical interest in the period 30-90 days after RC in a surgical hospital working according to the protocol for early postoperative recovery of the patient
Event-free survival | 90 days after Radical cystectomy
  Estimate the time to development of events of clinical interest in the period 30-90 days after RC in a surgical hospital

SECONDARY OUTCOMES:
Emergence of resistant | 30-90 days after Radical cystectomy
  To assess the probability of occurrence of acquired carbapenemase against the background of prolonged antibiotic prophylaxis
All-cause mortality | 90 days after Radical cystectomy
  Establish the frequency of 30-day, 90-day all-cause mortality after RC in a surgical hospital working according to the protocol for early postoperative patient recovery

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Berkut, PhD, Principal Investigator — FSBI "N.N. Petrov NMRC of oncology" MH of Russian Federation
Locations (1):
- FSBI "N.N. Petrov NMRC of oncology" MH of Russian Federation, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berkut MV, Belyaev AM, Galunova TY, Tyapkin NI, Reva SA, Nosov AK. Prolonged 120-h meropenem antibiotic prophylaxis in radical cystectomy compared to 24h standard antibiotic prophylaxis: Final analysis of the randomized clinical trial. Arab J Urol. 2024 Jul 3;22(4):235-242. doi: 10.1080/20905998.2024.2373399. eCollection 2024. PMID 39355793